CLINICAL TRIAL: NCT02319746
Title: COGNITIVE BEHAVIORAL THERAPY PROGRAM TO FIRST-EPISODE PSYCHOSIS PATIENTS AND CANNABIS ABUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Itxaso Ortega Gonzalez, Itxsaso Gonzalez Ortega, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COG-CON
Record Dates: First submitted 2014-12-10; First posted 2014-12-18 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: First-episode Psychosis; Cannabis Abuse
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): The subjects of experimental group will receive a cognitive-behavioral treatment program specific for reduce cannabis use composed of 16 weekly sessions (one hour in duration), in addition to regular psychiatric review and pharmacological treatment. The group will consist of 6-8 subjects.
  Interventions: Behavioral: Cognitive-behavioral therapy program to first-episode psychosis patients and cannabis abuse
- Control group (Active Comparator): The control group will receive standard care for psychotic episodes which includes pharmacological treatment and psychoeducation, following the same format as the experimental group. 16 weekly sessions of psychoeducation (one hour in duration) will be conducted, in addition to regular psychiatric review and pharmacological treatment. Like the experimental group the group will consist of 6-8 subjects.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy program to first-episode psychosis patients and cannabis abuse — The intervention program is focused on reducing the cannabis use, improving awareness of illness, adherence to treatment, identification of prodromes, psychosocial functioning improvement and relapse prevention.
  Arms: Experimental group
Behavioral: Psychoeducation — The aim of psychoeducation is that the patient understands and be able to manage the disease providing the tools and skills to symptoms management, to avoid relapse and contribute to their wellbeing.
  Arms: Control group

SUMMARY:
General objective:

To assess the effectiveness of a treatment program specific for cannabis abuse (cognitive behavioral treatment + pharmacological treatment) compared to standard treatment (pharmacological treatment + psychoeducation) in patients with first episodes psychosis (FEP) cannabis users.

Design A multicenter single-blind randomized study with 1 year of follow-up. The effectiveness of a treatment program specific for cannabis abuse (cognitive behavioral treatment + pharmacological treatment) compared to standard treatment (pharmacological treatment + psychoeducation) in patients with first episodes psychosis (FEP) cannabis users will be assessed.

Patients will be randomly assigned to one of two treatments:

1. Experimental group (N=50): Cognitive-behavioral treatment specific for cannabis abuse + pharmacological treatment
2. Control group (N=50): standard treatment: psychoeducation + pharmacological treatment

ELIGIBILITY:
Inclusion Criteria:

1. - Having a first psychotic episode. DSM-IV-TR diagnosis of a psychotic disorder (i.e. schizophrenia, schizophreniform disorder, schizoaffective disorder, delusional disorder, bipolar disorder, atypical psychosis, brief psychotic disorder, or major depressive disorder with psychotic symptoms).
2. - Being a regular cannabis user according DSM-IV
3. -Being in remission from the first psychotic episode (not exceeding 5 years).

Exclusion Criteria:

1. Presenting organic brain pathology.
2. Presenting mental retardation according to DSM-IV criteria.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Cannabis use reduction in the follow-up | Baseline, 16 weeks (posttreatment), at 3 and 6 months and at one year of follow up.
  To assess whether cannabis focused psychological intervention is associated with a cannabis use reduction according to Europ-ASI scale compared to standard treatment
Improvement in the development of psychotic disorder | Baseline, 16 weeks (posttreatment), at 3 and 6 months and at one year of follow up
  To assess whether cannabis focused psychological intervention is associated with an improvement in the development of psychotic disorder (ie, reduction of symptoms and improvement of psychosocial functioning) compared with standard treatment at the end of treatment and at follow-up (at three and six months and one year of follow-up).
Changes in the components of the endogenous cannabinoid system | Baseline, 16 weeks (posttreatment), at 3 and 6 months and at one year of follow up
  To determine whether changes in the components of the endogenous cannabinoid system at systematic level are produced in FEP cannabis abusers.
Normalizing the possible alterations in the endogenous cannabinoid system | Baseline, 16 weeks (posttreatment), at 3 and 6 months and at one year of follow up
  To assess whether treatment program specific for cannabis abstinence is capable of normalizing the possible alterations in the endogenous cannabinoid system in patients that reduce the cannabis use.

SECONDARY OUTCOMES:
Decrease the number of cannabis users | Baseline, 16 weeks (posttreatment), at 3 and 6 months and at one year of follow up
  To determinate the number of patient who use cannabis in the follow-up in each group
Decrease of negative and positive psychotic symptoms | Baseline, 16 weeks (posttreatment), at 3 and 6 months and at one year of follow up
  To compare the decrease of negative and positive psychotic symptoms measured by Positive and Negative Syndrome Scale (PANSS), at post-treatment and follow-up.
Decrease of manic, depressive and anxiety symptoms | Baseline, 16 weeks (posttreatment), at 3 and 6 months and at one year of follow up
  To compare the decrease of manic, depressive and anxiety symptoms at post-treatment and follow-up. Manic symptoms will be measured using Young Mania Rating Scale (YMRS). Anxiety and depressive symptoms will be measured using Hamilton Anxiety Scale (HAM-A) and Hamilton Depression Scale (HAM-D), respectively.
Improvement in the psychosocial functioning | Baseline, 16 weeks (posttreatment), at 3 and 6 months and at one year of follow up
  To compare the improvement of psychosocial functioning in each group by Functioning Assessment Short Test (FAST).
Improvement in the adherence to pharmacological treatment | Baseline, 16 weeks (posttreatment), at 3 and 6 months and at one year of follow up
  To compare the adherence to pharmacological treatment in each group using Morisky-Green Scale.
Withdrawal of patients | Baseline, 16 weeks (posttreatment), at 3 and 6 months and at one year of follow up
  To evaluate percentage of withdrawal in the follow-up.
Decrease the number of relapses and rehospitalizations | Baseline, 16 weeks (posttreatment), at 3 and 6 months and at one year of follow up
  To compare the number of relapses and rehospitalizations in in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Araba University Hospital, Vitoria-Gasteiz, Alava, Spain

REFERENCES:
- [Derived] Gonzalez-Ortega I, Echeburua E, Garcia-Alocen A, Vega P, Gonzalez-Pinto A. Cognitive behavioral therapy program for cannabis use cessation in first-episode psychosis patients: study protocol for a randomized controlled trial. Trials. 2016 Jul 29;17:372. doi: 10.1186/s13063-016-1507-x. PMID 27473688